CLINICAL TRIAL: NCT05419778
Title: Clinical Evaluation Of Soft Tissue Closure In Alveolar Ridge Preservation Procedures
Brief Title: Alveolar Ridge Preservation Procedures
Status: Completed | Type: Observational
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: 18-06428-FB
Record Dates: First submitted 2022-05-16; First posted 2022-06-15 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-05

CONDITIONS: Alveolar Ridge Preservation
Keywords: Bone; OsteoGen; Cortico-Cancellous; Foreign body reaction
MeSH Terms: conditions — Foreign-Body Reaction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Excess tissue will be collected if the subject has a standard of care implant-related procedure where tissue could need to be removed for implant placement purposes. For example, if a patient undergoes a tooth extraction, ridge augmentation, and implant placement then any portion of the excised tooth and connective tissue will be kept for later analyses of histology discovery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A (Osteogen plug®): The surgical procedure will be conducted following standard procedures for tooth exodontia and ridge preservation. The selected individual sites will be subjected to the standard of care extraction protocol and then randomized to receive treatment with a type I bovine Achilles tendon collagen with bioactive resorbable calcium apatite crystals (CCAC)(Osteogen) ridge augmentation procedures. Intra-oral photographs will be made at the same optic focal distance using a ruler which will be used to evaluate areas where the membrane is still exposed and not epithelized. At 4-6 weeks and again at 20 weeks postoperatively, each study subject will return for implant placement in the ridge preservation area.
  Interventions: Device: Osteogen plug®
- Group B ( MInerOss® ): The surgical procedure will be conducted following standard procedures for tooth exodontia and ridge preservation. The selected individual sites will be subjected to the standard of care extraction protocol and then randomized to a cortico-cancellous bone chips mix with polytetrafluoroethylene (dPTFE)(Cytoplast) barrier membrane ridge augmentation procedures. Intra-oral photographs will be made at the same optic focal distance using a ruler which will be used to evaluate areas where the membrane is still exposed and not epithelized. At 4-6 weeks and again at 20 weeks postoperatively, each study subject will return for implant placement in the ridge preservation area.
  Interventions: Device: MInerOss®

INTERVENTIONS:
Device: Osteogen plug® — A type I bovine Achilles tendon collagen with bioactive resorbable calcium apatite crystals (CCAC)
  Groups: Group A (Osteogen plug®)
Device: MInerOss® — A cortico-cancellous bone chips mix with polytetrafluoroethylene (dPTFE)(Cytoplast) barrier membrane.
  Groups: Group B ( MInerOss® )

SUMMARY:
Tooth loss is accompanied by different patterns of bone loss. Up to 50% loss of alveolar crestal bone width will likely occur 1 year after tooth loss, especially in the anterior maxilla. A great percentage of the process of alveolar bone resorption occurs within the first 3 to 6 months post-extraction. If ridge preservation is not conducted, 40%-60% of the total alveolar bone volume is lost during the first 2-3 years post-extraction, and this phenomenon has shown to continue to occur at a rate of 0.25%-0.5% loss per year. It has been proposed that ridge augmentation procedures may reduce the expected ridge reduction after tooth loss. Ridge augmentation procedures may require the use of bone grafts and non-resorbable or non-resorbable barrier membranes. The use of non-resorbable barrier membranes for ridge augmentation has the clinical disadvantage of needing a second procedure for its removal during the healing phase. Osteogen® plug (OPP) consists of a non-ceramic bone graft incorporated in type I bovine Achilles tendon collagen. OPP was first developed to serve as a one-step grafting solution for ridge preservation without the need for a barrier membrane

DETAILED DESCRIPTION:
There will be two(2) groups of standardized treatment (tooth extractions will not take place for research purposes. The Periodontal clinic receives referred tooth extraction indications for treatment as part of the patient's overall treatment plan) evaluated for this study. Subjects will be randomized to either treatment a) standard of care treatment for tooth extraction and ridge augmentation procedures with Cytoplast GRB, or b) standard of the care treatment protocol and ridge augmentation procedures with Osteogen.

Each individual extraction site of the enrolled subject will be randomly assigned to Group A and/or Group B for the ridge augmentation procedure. It is possible for a subject to be randomized to both treatment groups. Randomization is like a "coin toss" prior to the initiation of the surgical procedure. The "coin toss" will be to define the procedure to be conducted for the smallest tooth number first. A computer-generated randomization assignment has been populated for the ridge augmentation assignments. The surgical procedure will be conducted following standard procedures for tooth exodontia and ridge preservation.The selected individual sites will be subjected to the standard of care extraction protocol and then randomized to one of two(2) ridge augmentation procedures. Intra-oral photographs will be made at the same optic focal distance using a ruler which will be used to evaluate areas where the membrane is still exposed and not epithelized. At 20 weeks postoperatively, each study subject will return for implant placement in the ridge preservation area. Excess tissue will be collected if the subject has a standard of care implant-related procedure where tissue could need to be removed for implant placement purposes. For example, if a patient undergoes a tooth extraction, ridge augmentation, and implant placement then any portion of the excised tooth and connective tissue will be kept for later analyses of histology discovery. No additional tissue will be collected for research purposes. There will be one screening visit, a treatment visit, and 7 post-operative follow-up visits at 1, 2, 3, 4, 6, 8, and 20 weeks. Subjects will visit the clinic a total of eight (9) times. Of the 9 visits, 1 visit is standard of care, 3 visits are a combined standard of care and research procedure visits and 5 are strictly for research purposes. The nonabsorbable membranes in the control will be removed after 4-6 weeks in a most atraumatic manner with the help of a tweezer without disturbing the underlying new connective tissue formation. As there is no need for removal of the absorbable membrane in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* UT Clinic Participates

  * Participates that live within 100 miles of UTHSC.
  * Participates at least 12 years of age. If participants are 13-14 years of age, the premolars and molars will be included in this study. #2-15 & #18-31.
  * Participates willing to cooperate with the post-operative instructions;
  * Participates with 2 or more (multiples of 2) teeth needing Maxillary/mandibular and anterior/posterior teeth extractions without restrictions due to the percentage of surface area after the extraction and not interfering with the tooth's alveolar soft tissue exposed surface area.
  * Participates with the availability of returning for 8 visits for data collection.
  * Participants are willing to cooperate with answering the VAS and taking standardized photographs.
  * Participants are physically able to tolerate surgical procedures based on current medical history.
  * Participates able to provide voluntary consent; read and understand English

Exclusion Criteria:

* Participates with Diabetes
* History of use of bisphosphonates
* Current smoker
* If the participant is 12-13 years of age, the tooth/teeth to be removed will not be a primary tooth due to the permanent teeth developing underneath the primary teeth.
* Pregnant and lactating women

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Up to twenty (20) participants, at least 12 years old, needing a tooth (teeth) extraction(s) with a combined extraction site preservation treatment of 20 extraction sites.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Histological Bone Formation Changes | 4 weeks
  histomorphometric evaluation of the grafted bone. The area fraction (AF) of newly formed bone was measured automatically. The area fraction represents the percentage of the newly formed bone trabeculae to the total area of the microscopic field. The mean area fraction (MAF) for each case was calculated. Estimation of osteocytes count in each microscopic field, viable osteocytes within their lacunae in the newly formed bone
Histological Bone Formation Changes | 6 weeks
  histomorphometric evaluation of the grafted bone. The area fraction (AF) of newly formed bone was measured automatically. The area fraction represents the percentage of the newly formed bone trabeculae to the total area of the microscopic field. The mean area fraction (MAF) for each case was calculated. Estimation of osteocytes count in each microscopic field, viable osteocytes within their lacunae in the newly formed bone
Histological Bone Formation Changes | 20 weeks
  histomorphometric evaluation of the grafted bone. The area fraction (AF) of newly formed bone was measured automatically. The area fraction represents the percentage of the newly formed bone trabeculae to the total area of the microscopic field. The mean area fraction (MAF) for each case was calculated. Estimation of osteocytes count in each microscopic field, viable osteocytes within their lacunae in the newly formed bone
Clinical Dimensional Changes | 4 weeks
  * Clinical evaluation of alveolar ridge bucco-lingually dimensional changes following alveolar ridge augmentation using standardized photography.
  * Clinical evaluation of alveolar ridge bucco-lingually dimensional changes following alveolar ridge augmentation using digital planimetry program, SigmaScan Pro 5.0.
Clinical Dimensional Changes | 6 weeks
  * Clinical evaluation of alveolar ridge bucco-lingually dimensional changes following alveolar ridge augmentation using standardized photography.
  * Clinical evaluation of alveolar ridge bucco-lingually dimensional changes following alveolar ridge augmentation using digital planimetry program, SigmaScan Pro 5.0.
Clinical Dimensional Changes | 20 weeks
  * Clinical evaluation of alveolar ridge bucco-lingually dimensional changes following alveolar ridge augmentation using standardized photography.
  * Clinical evaluation of alveolar ridge bucco-lingually dimensional changes following alveolar ridge augmentation using digital planimetry program, SigmaScan Pro 5.0.
Evaluate Patient Pain | 20 weeks
  Evaluate patient pain during the wound healing phase using the visual analog scale (VAS).
  Scale range (0-10) : 0 1 2 3 4 5 6 7 8 9 10 Minimum Value: 0 = no pain Maximum Value: 10 = worse pain ever imaged

CONTACTS AND LOCATIONS:
Overall Officials: Cimara F Ferreira, PhD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

REFERENCES:
- [Background] Molnar JA, Lew WK, Rapp DA, Gordon ES, Voignier D, Rushing S, Willner W. Use of standardized, quantitative digital photography in a multicenter Web-based study. Eplasty. 2009;9:e4. Epub 2009 Jan 12. PMID 19212431
- [Background] McCormack HM, Horne DJ, Sheather S. Clinical applications of visual analogue scales: a critical review. Psychol Med. 1988 Nov;18(4):1007-19. doi: 10.1017/s0033291700009934. PMID 3078045
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Nevins M, Camelo M, De Paoli S, Friedland B, Schenk RK, Parma-Benfenati S, Simion M, Tinti C, Wagenberg B. A study of the fate of the buccal wall of extraction sockets of teeth with prominent roots. Int J Periodontics Restorative Dent. 2006 Feb;26(1):19-29. PMID 16515093
- [Background] Tallgren A. The continuing reduction of the residual alveolar ridges in complete denture wearers: a mixed-longitudinal study covering 25 years. 1972. J Prosthet Dent. 2003 May;89(5):427-35. doi: 10.1016/s0022-3913(03)00158-6. No abstract available. PMID 12806317
- [Background] Ashman A. Postextraction ridge preservation using a synthetic alloplast. Implant Dent. 2000;9(2):168-76. doi: 10.1097/00008505-200009020-00011. PMID 11307396
- [Background] Fickl S, Schneider D, Zuhr O, Hinze M, Ender A, Jung RE, Hurzeler MB. Dimensional changes of the ridge contour after socket preservation and buccal overbuilding: an animal study. J Clin Periodontol. 2009 May;36(5):442-8. doi: 10.1111/j.1600-051X.2009.01381.x. PMID 19419446
- [Background] Barber HD, Lignelli J, Smith BM, Bartee BK. Using a dense PTFE membrane without primary closure to achieve bone and tissue regeneration. J Oral Maxillofac Surg. 2007 Apr;65(4):748-52. doi: 10.1016/j.joms.2006.10.042. PMID 17368373
- [Background] Lekovic V, Camargo PM, Klokkevold PR, Weinlaender M, Kenney EB, Dimitrijevic B, Nedic M. Preservation of alveolar bone in extraction sockets using bioabsorbable membranes. J Periodontol. 1998 Sep;69(9):1044-9. doi: 10.1902/jop.1998.69.9.1044. PMID 9776033
- [Background] Wang HL, Boyapati L. "PASS" principles for predictable bone regeneration. Implant Dent. 2006 Mar;15(1):8-17. doi: 10.1097/01.id.0000204762.39826.0f. PMID 16569956
- [Background] Kosinski T. A Simple and Cost-Effective Socket Preservation Technique. Dent Today. 2016 Apr;35(4):90, 92, 94-5. No abstract available. PMID 27244995
- [Background] Feng L, Zhang L, Cui Y, Song TX, Qiu ZY, Wang XM, Tan BS. Clinical evaluations of mineralized collagen in the extraction sites preservation. Regen Biomater. 2016 Mar;3(1):41-8. doi: 10.1093/rb/rbv027. Epub 2016 Jan 19. PMID 26815224
- [Background] Nevins M, Parma-Benfenati S, Janke UW, Kleyer A, Rasperini G, Tinti C, Schupbach P, Kim DM. The efficacy of mineralized allograft cortical and cancellous chips in maxillary sinus augmentations. Int J Periodontics Restorative Dent. 2014 Nov-Dec;34(6):789-93. doi: 10.11607/prd.1720. PMID 25411734
- [Background] Park JC, Koo KT, Lim HC. The hidden X suture: a technical note on a novel suture technique for alveolar ridge preservation. J Periodontal Implant Sci. 2016 Dec;46(6):415-425. doi: 10.5051/jpis.2016.46.6.415. Epub 2016 Dec 26. PMID 28050319
- [Result] Evian CI, Rosenberg ES, Coslet JG, Corn H. The osteogenic activity of bone removed from healing extraction sockets in humans. J Periodontol. 1982 Feb;53(2):81-5. doi: 10.1902/jop.1982.53.2.81. PMID 6950085
- [Result] Dahlin C, Linde A, Gottlow J, Nyman S. Healing of bone defects by guided tissue regeneration. Plast Reconstr Surg. 1988 May;81(5):672-6. doi: 10.1097/00006534-198805000-00004. PMID 3362985
- [Result] Beth-Tasdogan NH, Mayer B, Hussein H, Zolk O. Interventions for managing medication-related osteonecrosis of the jaw. Cochrane Database Syst Rev. 2017 Oct 6;10(10):CD012432. doi: 10.1002/14651858.CD012432.pub2. PMID 28983908

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT05419778/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT05419778/ICF_001.pdf